CLINICAL TRIAL: NCT03460015
Title: Evaluation of Sevoflurane in Chronic Obstructive Pulmonary Disease Exacerbation in Intensive Care Unit: A Comparative Prospective Study
Brief Title: Sevoflurane in Chronic Obstructive Pulmonary Disease Exacerbation
Acronym: SEVOCOPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention The study was terminated prematurely due to inclusion difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9856
Record Dates: First submitted 2018-02-01; First posted 2018-03-09 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: COPD Exacerbation; Invasive Mechanical Ventilation
Keywords: COPD exacerbation; Sevoflurane; Airway Resistance
MeSH Terms: interventions — Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Experimental)
  Interventions: Drug: Sevoflurane; Drug: Propofol
- Propofol group (Active Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — During the first 30 minutes after randomization, patients will be treated with propofol (same dosage as the propofol group).
  Once the AnaConDa® system is installed, sevoflurane administration will begin (propofol is stopped).
  Arms: Sevoflurane group
Drug: Propofol — In the control group, sedation will be maintained with the above objective (RASS between -4 and -5, BIS between 40 and 60) until the patient is extubated.
  In the sevoflurane group, propofol is administrated during the first 30 minutes after the randomization and when the AnaConDa® system is installed propofol is stopped.

SUMMARY:
Prospective, open-label, single-center, study to investigate the effect of sevoflurane sedation compared to a propofol-controlled arm during COPD exacerbation requiring invasive mechanical ventilation in ICU.

Primary outcome measure:

Evolution of airway resistance before and after sevoflurane in COPD patients,

Secondary outcomes measures:

Respiratory mechanics (Maximum pressure, PEEPi and PEEPtot, trapped volume), Gas exchange by the help of blood gases, The heterogeneity of alveolar ventilation by electro-impedancemetry, Evolution of pulmonary inflammation, Trophicity and contractility of the diaphragm,

ELIGIBILITY:
Inclusion Criteria :

* COPD exacerbation
* Invasive mechanical ventilation and sedation for a planned duration of at least 24 hours
* Consent
* Age ≥ 18 years
* Affiliation or beneficiary of a social security scheme

Exclusion Criteria :

* Contraindication to the administration of sevoflurane (personal or family history of malignant hyperthermia, allergy or halogenated anesthetic accident, chronic myopathy, halogenated toxic hepatitis, uncontrolled intracranial hypertension, unexplained leukocytosis after anesthesia with a halogenated agent)
* Contraindication to the administration of propofol (known hypersensitivity to propofol, soy, peanut or any of the excipients of the emulsion, antecedent of Propofol Related Infusion Syndrome)
* Refusal of consent
* Guardianship
* Age < 18 years
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Evolution of airway resistance before and after sevoflurane in COPD patients | Hour 48
  Total airway resistance will be measured using the ventilator by setting a 5s inspiratory pause and to measure the sum of (Pmax-P1)/Flow + (P1-Pplat)/Flow. The mechanical ventilation setting will be standardised during the study period and will be similar between the two groups.

SECONDARY OUTCOMES:
Maximum pressure | Evolution between Hour 0 and Hour 48
PEEPi | Evolution between Hour 0 and Hour 48
PEEPtot | Evolution between Hour 0 and Hour 48
Trapped volume | Evolution between Hour 0 and Hour 48
Gas exchange by the help of blood gases | Evolution between Hour 0 and Hour 48
Heterogeneity of alveolar ventilation by electro-impedancemetry | Evolution between Hour 0 and Hour 48
Proinflammatory cytokines (IL1, IL6, TNFalpha) and sRAGE measurements in miniBroncho-Alveolar lavages | Evolution between Hour 0 and Hour 48
Thickness of the diaphragm measured by ultrasound | Evolution between Hour 0 and Hour 48

CONTACTS AND LOCATIONS:
Overall Officials: Boris Jung, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, Hérault, France